CLINICAL TRIAL: NCT02069275
Title: Patients Immediate Mobilization After Coronary Angiography and Percutaneous Coronary Intervention. Is it SAfe to MObilize Patients Very eARly After Cardiac Catheterisation?
Brief Title: Immediate Mobilization After Cardiac Catheterisation
Acronym: SAMOVAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marianne Wetendorff Noergaard, Clinical Nurse Specialist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SAMOVAR 01
Record Dates: First submitted 2014-02-13; First posted 2014-02-24 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Vascular Access Complication; Comfort
Keywords: Immediate mobilization; Bedrest; Coronary angiography; Coronary percutaneous intervention; Vascular access complications; Patients comfort
MeSH Terms: interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate mobilization (Experimental): Immediate mobilization after coronary angiography or percutaneous coronary intervention
  Interventions: Other: Immediate mobilization
- Two hours bedrest (Active Comparator): Bedrest two hours after coronary angiography or percutaneous coronary intervention
  Interventions: Other: Two hours bedrest

INTERVENTIONS:
Other: Immediate mobilization — Patients are mobilized immediate after coronary angiography and percutaneous coronary intervention via femoral access and closed with Angio-seal closing device. Heparin reverted with Protaminsulphate
  Arms: Immediate mobilization
Other: Two hours bedrest — Patients is following the usual regimen, two hours bedrest after coronary angiography and percutaneous coronary intervention via femoral access and closed with Angio-seal closing device before mobilization. Heparin is reverted with Protaminsulphate
  Arms: Two hours bedrest

SUMMARY:
The purpose of this study is to investigate the frequency of bleeding and haematomas in patients undergoing coronary angiography or percutaneous coronary intervention via femoral artery and mobilized immediately after the procedure, compared to those mobilized after two hours (following the standard regimen). At the same time the investigators will investigate whether it reduces the discomfort being mobilized immediately after the procedure.

DETAILED DESCRIPTION:
The frequency of hematoma, bleeding or pseudoaneurysm at the access site in the groin is 7-15% with regimens that involve 0-2 hours of bed rest, somewhat more frequent after Percutaneous coronary intervention (PCI) than coronary angiography (CAG). There seems to be no reduction in the complications of the CAG or PCI by maintaining the bed rest for more than 2 hours after the procedure. Angio-Seal seems most effective of current closure devices. There is less discomfort associated with early compared with late mobilization. Protamine reverse heparin's effect without the side effects of that regime.

There lacks a larger randomized study of the safety of mobilizing patients immediately after CAG and after PCI.

ELIGIBILITY:
Inclusion Criteria:

* CAG or PCI performed via the femoral artery
* No hematoma in the groin (> 5 cm in diameter)
* Heparin reversed with protamine after PCI

Exclusion Criteria:

* Oozing, bleeding or hematoma
* Treatment with Integrilin, ReoPro, or Marevan
* Heparin can not be reversed
* The patient does not want to participate
* Systolic blood pressure > 180 mm Hg after the procedure
* BMI> 35 (can be modified if the groin can be assessed in an upright position)
* Demented, unconscious patients who do not understand the information for participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Hematoma> 5 cm | participants will be followed for the duration of hospital stay, an expected average of 24 hours
  occurred after the end of the procedure, including retroperitoneal hematoma, bleeding requiring transfusion or pseudoaneurysm that require vascular surgical intervention. Assessed after 30 minutes, after two hours and before discharge

SECONDARY OUTCOMES:
The presence of hematoma> 10 cm in diameter | participants will be followed for the duration of hospital stay, an expected average of 24 hours
The presence of hematoma 2-5 cm in diameter | participants will be followed for the duration of hospital stay, an expected average of 24 hours
Oozing or bleeding from the puncture site | participants will be followed for the duration of hospital stay, an expected average of 24 hours
Comfort rating (NRS scale) | Two hours after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marianne W Moergaard, MVO, Principal Investigator — Cardiac Cath.lab. Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Norgaard MW, Faerch J, Joshi FR, Hofsten DE, Engstrom T, Kelbaek H. Is It Safe to Mobilize Patients Very Early After Transfemoral Coronary Procedures? (SAMOVAR): A Randomized Clinical Trial. J Cardiovasc Nurs. 2022 Sep-Oct 01;37(5):E114-E121. doi: 10.1097/JCN.0000000000000845. Epub 2021 Jul 26. PMID 34321432